CLINICAL TRIAL: NCT05450393
Title: Prospective Collection of PillCamTM SB3 Capsule Endoscopy and Device-Assisted Enteroscopy Procedures Data for Development of an Artificial Intelligence Software System to Apply to Endoscopy Procedures (GPS Study)
Brief Title: Data Collection of PillCamTM SB3 Capsule Endoscopy and Device-Assisted Enteroscopy Routine Care Procedures (GPS Study)
Status: Withdrawn | Type: Observational
Why Stopped: Study was cancelled by sponsor due to priority realignment
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT21042
Record Dates: First submitted 2022-06-28; First posted 2022-07-08 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2023-10

CONDITIONS: Small Intestine Disease; Small Intestine Cancer; Small Intestinal Ulcer Bleeding; Small Intestine Obstruction; Small Intestine Adenocarcinoma; Small Intestine Polyp

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PillCam SB procedure and deep enteroscopy (Device-assisted enteroscopy, DAE): Subjects with abnormal PillCam SB3 procedure followed by DAE (if performed).

SUMMARY:
A prospective, multicenter, post-market, minimal risk, observational study designed to collect PillCamTM SB3 capsule endoscopy (CE) procedures and subsequent device-assisted enteroscopy (DAE) procedures data (double balloon enteroscopy (DBE), single balloon enteroscopy (SBE) and spiral enteroscopy (SE)) in medical centers in the United States (US).

DETAILED DESCRIPTION:
A prospective, multicenter, post-market, minimal risk, observational study designed to collect up to 60 PillCamTM SB3 CE procedures and subsequent DAE procedures data (double balloon enteroscopy (DBE), single balloon enteroscopy (SBE) and spiral enteroscopy (SE)) in up to 6 medical centers in the United States (US). The data will be collected from subjects who underwent standard of care (SOC) PillCamTM SB3 CE procedure and were referred to a subsequent SOC DAE. In addition, relevant surgical, endoscopic and histology reports as well as radiological data (such as CT, Magnetic Resonance Enterography (MRE) images and reports) may be collected retrospectively 6 months prior to enrollment and prospectively 3 months post enrollment, when applicable. In addition, up to 400 PillCamTM SB3 CE procedures data may be collected from subjects who underwent SB3 procedure (not necessarily followed by DAE) and abnormal SB findings were indicated in their CE report. Study duration is up to 3 years from initial Institutional Review Board (IRB) approval.

Collected data will include PillCamTM raw data, videos and reports, as well as DAE reports, videos and histology reports (when applicable). Demographic data will also be collected to provide a description of the study population characteristics and disposition. All the collected data will be de-identified by delegated and authorized sites' team members, in a manner that is untraceable by the sponsor. The data will be used by Medtronic Gastrointestinal research and development (R&D) team in collaboration with third parties, including but not limited to external physicians and R&D partners, as applicable, for development of an Artificial Intelligence (AI) software system to apply to endoscopy procedures, as well as for SB pathologies detection development and validation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects (≥18 years)
2. The subject underwent a SOC PillCamTM SB3 CE procedure and is referred to a subsequent DAE procedure(s), as part of the routine care or The subject underwent a SOC PillCamTM SB3 CE procedure (not necessarily followed by a DAE) and abnormal findings were indicated in the CE report (optional).
3. The subject received an explanation and understands the nature of the study and provided oral consent.

Exclusion Criteria:

1. The subject is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent standard of care (SOC) PillCamTM SB3 CE and subsequent DAE procedures or Subjects who underwent SOC PillCamTM SB3 CE procedures only and abnormal findings were indicated in their CE report (optional).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Prospective collection of PillCamTM SB3 capsule endoscopy and DAE procedures data | Up to 3 years from study approval
  Collection of GI pathologies data along with descriptive demographics data for research and development purposes.

IPD SHARING:
Plan to Share IPD: No